CLINICAL TRIAL: NCT01398189
Title: Validation of Molecular Imaging Technologies for Early Clinical Trials
Brief Title: F-18 Altanserin PET Study of Patients Receiving Clozapine
Acronym: APC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae Seung Chang, Clinical Assistant Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SNUBH 04-2011-050
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: clozapine; PET; schizophrenia; schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- clozapine (Experimental): patients with refractory schizophrenia or schizoaffective disorder
  Interventions: Drug: clozapine

INTERVENTIONS:
Drug: clozapine — C-11 clozapine
  Other Names: clozaril

SUMMARY:
To examine the feasibility of molecular imaging markers in clinical psychopharmacology

DETAILED DESCRIPTION:
Clinical evaluation of patients with psychiatric disorders is mainly dependent on patients' reports and clinicians' observations. In order to develop objective and quantifiable measures of psychopathology, molecular imaging techniques will be used in patients receiving clozapine.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males as determined by medical history and physical examination
* Age from 19 to 45 years
* Weight ≥ 45 kg and within ± 20% of IBW
* Clinical laboratory test results within normal reference range for the National Cancer Center, Hospital or results with minor deviations which are judged to be not clinically significant by the investigator
* Normal blood pressure and heart rate (supine and standing) as determined by the investigator
* Are reliable and willing to make themselves available for the duration of the study, and who will abide by the study restrictions
* Have given written informed consent

Exclusion Criteria:

* Evidence of significant active hematologic disease
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neurological disorders capable of altering the absorption, metabolism or elimination of drugs, or of constituting a risk factor when taking the study medication
* An episode of febrile disease or infectious disease within the past 2 weeks
* Evidence of significant active neuropsychiatric disease
* Regular use of drugs or abuse
* History of drug hypersensitivity or clinically significant allergic reactions of any origin
* Participation in a study involving administration of an investigational compound within the past 30 days
* Use of any current medication
* Smoking history for recent 3 months

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
pharmacodynamics of F-18 artanserin | 84 days
  PET imaging with F-18 altanserin infusion

SECONDARY OUTCOMES:
serum level of clozapine and metabolites | 84 days
  dose-response relationship between clozapine and receptor occupancy

CONTACTS AND LOCATIONS:
Overall Officials: Jae Seung Chang, MD, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea